CLINICAL TRIAL: NCT05561699
Title: Sequential Preoperative Penpulimab Combined With Chemoradiotherapy(CRT) for Locally Advanced Esophageal Squamous Cell Cancer: A Prospective, Single Arm, Single Center，Exploratory Study
Brief Title: Sequential Preoperative Penpulimab Combined With Chemoradiotherapy(CRT) for Locally Advanced Esophageal Squamous Cell Cancer
Acronym: SPEED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2022-143R2
Record Dates: First submitted 2022-09-28; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Penpulimab Combined With Chemoradiotherapy(CRT) (Experimental)
  Interventions: Drug: Penpulimab Combined With CRT

INTERVENTIONS:
Drug: Penpulimab Combined With CRT — 1. Penpulimab: 200mg, intravenous infusion, once every two weeks. After completing two courses of CRT, continue to send Penpulimab 200mg every two weeks on the first and 14th days after the completion of CRT, two courses of treatment, a total of four courses.
  2. Radiotherapy 40gy/20fx, once a day from Monday to Friday, completed in 4 weeks;
  3. PC regimen: Paclitaxel 50mg/m2, intravenous drip, carboplatin AUC=2mg/ml/min, intravenous drip, once a week during radiotherapy, a total of 4 courses, the specific time is D1, 8, 15, 22 days after the beginning of radiotherapy.
  4. Gastrointestinal reactions such as nausea and vomiting should be routinely prevented before chemotherapy. Dexamethasone 10mg should be used 30 ~ 60 minutes before paclitaxel, and intramuscular injection should be stopped immediately in case of drug or infusion reactions.

SUMMARY:
This study used an open single center study design to observe the efficacy and safety of Penpulimab combined with Chemoradiotherapy(CRT) in preoperative T2,3,4aN0-1-2M0 esophageal squamous cell carcinoma (ESCC).

ELIGIBILITY:
Inclusion Criteria:

* Resectable t2,3,4an0-1-2m0 esophageal squamous cell carcinoma initially diagnosed by histology or cytology;
* Without any systematic anti-tumor treatment;
* ECOG 0-1;
* ANC≥ 1.5×109/L;
* PLT≥ 75×109/L;
* HB≥ 8.0 g/dL;
* TBIL ≤ 1.5´ ULN;
* ALT and AST ≤ 2.5´ULN;
* Cr ≤ 1.5´ULN or CCr ≥ 60ml/min;
* Urine protein < +, if urine protein + then the total protein in 24 hours must be <500mg;
* Blood glucose is within the normal range and / or patients with diabetes are in treatment, but blood glucose is controlled in a stable state;
* FEV1 ≥ 2L; If the baseline FEV1 is less than 2L, it is estimated that the FEV1 after surgery is greater than 800ml；
* No myocardial infarction within 1 year; No unstable angina pectoris; No symptomatic severe arrhythmia; No cardiac insufficiency；
* There are no serious complications or other major diseases that have not been cured；
* Thoracic surgeons judge those who can tolerate the operation；
* Female subjects with fertility and male subjects with partners of childbearing age need to use a medically approved contraceptive measure during the study treatment and at least 6 months after the last chemotherapy；
* The subjects voluntarily joined the study and signed the informed consent form

Exclusion Criteria:

* Received any kind of systematic anti-tumor treatment before the first use of the study drug；
* At the same time, another clinical study will be included, unless it is an observational (non intervention) clinical study；
* Subjects who need to be given corticosteroids (more than 10mg prednisone equivalent dose per day) or other immunosuppressants for systematic treatment within 2 weeks before the first use of the study drug；
* Have been vaccinated with tumor vaccine or have been vaccinated with live vaccine within 4 weeks before administration；
* Have a history of active autoimmune diseases and autoimmune diseases; Except for patients who have recovered from childhood asthma / allergy and do not need any intervention after adulthood; Autoimmune mediated hypothyroidism treated with a stable dose of thyroid hormone replacement; Use a stable dose of insulin for type I diabetes；
* Serious interference occurred within 4 weeks before the first use of the study drug (CTC AE>2); Baseline chest imaging examination showed active pulmonary inflammation, symptoms and signs of infection within 2 weeks before the first use of the study drug, or the need for oral or intravenous antibiotics；
* Have a history of interstitial lung disease；
* The subjects had active hepatitis B (HBV DNA ≥ 2000 IU/ml or 104copies/ml), hepatitis C (hepatitis C antibody positive and HCV-RNA higher than the lower limit of the analysis method);
* Pregnant or lactating women;
* There are serious complications or other major diseases that have not been cured;
* Patients judged by thoracic surgeons to be intolerant of surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-09-28 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
pathological complete remission（pCR）rate | 3 to 4 months
  Proportion of subjects who achieved pathological complete remission (PCR)，PCR was defined as the microscopic absence of tumor cells in the pathological evaluation of excised esophageal cancer lesions and regional lymph node samples after surgery.
safety（AE or SAE） | 2 to 3 years from baseline
  Incidence of adverse events or serious adverse events

SECONDARY OUTCOMES:
Tumor regression grade（TRG） | 3 to 4 months
  Evaluation of the focus of primary tumor after radiotherapy and chemotherapy
R0 resection rate | 3 to 4 months
  Proportion of subjects reaching R0 resection. resection was defined as no tumor cells remained within 1mm of the two cutting edges of the esophageal cancer lesions removed during the operation.
Event free survival（EFS） | 2 to 3 years from baseline
  Date of first administration to date of first recording of relevant events
Overall survival（OS） | 2 to 3 years from baseline
  Date of first administration to date of death due to any cause
Disease free survival（DFS） | 2 to 3 years from baseline
  Date from the operation to the first recording of relevant events

CONTACTS AND LOCATIONS:
Overall Officials: Jian Wang, MD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China